CLINICAL TRIAL: NCT02146612
Title: An Observational Study to Evaluate Amino Acid Usage Patterns in Daily Practice
Brief Title: Amino Acid Usage Patterns in Daily Practice
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: ANTK1202
Record Dates: First submitted 2014-04-24; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Wounds; Lean Body Mass
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group Receiving Supplement: Amino acid supplement group
  Interventions: Other: Amino Acid Supplement Group

INTERVENTIONS:
Other: Amino Acid Supplement Group — Group receiving nutritional supplement

SUMMARY:
The present study aims to evaluate the patient profile including medical conditions who use a nutritional supplement along with a balanced and varied diet in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Consuming amino acid containing oral nutritional supplement before enrolment for malnutrition for hard-to-heal wounds or malnutrition due to primary disease.
* Followed by internal medicine or surgery departments.

Exclusion Criteria:

* History of allergy or hypersensitive reaction to any ingredient in the amino acid containing oral nutritional supplement.
* History of any food allergy or intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects receiving amino acid supplement prior to enrollment
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Frequencies of Medical Conditions | Baseline
  Diagnosis information

SECONDARY OUTCOMES:
Intake of Amino Acid containing Nutrition Supplement | Baseline and Week 8
Anthropometrics | Change from Baseline to Week 8
  weight, BMI
Laboratory Parameters | Change from Baseline to Week 8
  Pre-albumin/Albumin

CONTACTS AND LOCATIONS:
Overall Officials: Tahsin Ozcagli, MD, Study Chair — Abbott Nutrition Turkey
Locations (18):
- Turkey (Türkiye) (18):
  - Adana Numune Eğitim ve Araştırma Hastanesi, Adana
  - Çukurova Üniversitesi Tıp Fakültesi, Adana
  - ANKARA ATATÜRK Eğitim ve Araştırma Hastanesi, Ankara
  - Ankara Numune Eğitim ve Araştırma Hastanesi, Ankara
  - Dışkapı Yıldırım Beyazıt Eğitim ve Araştırma Hastanesi, Ankara
  - Gazi Üniversitesi Tıp Fakültesi, Ankara
  - Bursa Çekirge Devlet Hastanesi, Bursa
  - Uludağ Üniversitesi Tıp Fakültesi, Bursa
  - Acıbadem Eskişehir Hospital, Eskişehir
  - Fatih Sultan Mehmet Eğitim ve Araştırma Hastanesi, Istanbul
  - GÜLHANE ASKERİ TIP AKADEMİSİ - İstanbul, Istanbul
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi, Istanbul
  - T.C.Bezmiâlem Vakıf Üniversitesi Tıp Fakültesi Hastanesi, Istanbul
  - Dr. Suat Seren Gogus Hastaliklari Hastanesi, Izmir
  - Ege Üniversitesi Tıp Fakültesi, Izmir
  - Erciyes Üniversitesi Tıp Fakültesi, Kayseri
  - Ondokuz Mayıs Üniversitesi Tıp Fakültesi, Samsun
  - Karadeniz Teknik Üniversitesi Tıp Fakültesi, Trabzon